CLINICAL TRIAL: NCT03259620
Title: A Phase 3, Randomized, Double-Blind, Vehicle-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of CLS006 Versus Vehicle in Subjects 2 Years of Age or Older With Cutaneous Common Warts
Brief Title: A Study to Evaluate the Safety and Efficacy of CLS006 Versus Vehicle in Subjects 2 Years of Age or Older With Cutaneous Common Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS006-CO-PR-002
Record Dates: First submitted 2017-08-22; First posted 2017-08-23 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Cutaneous Common Warts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLS006 (Experimental): Furosemide Topical Gel, 0.125%
  Interventions: Drug: CLS006
- CLS006 Vehicle (Experimental): Vehicle Topical Gel
  Interventions: Drug: CLS006 Vehicle

INTERVENTIONS:
Drug: CLS006 — Furosemide Topical Gel
  Arms: CLS006
Drug: CLS006 Vehicle — Vehicle Topical Gel
  Arms: CLS006 Vehicle

SUMMARY:
To evaluate the efficacy and safety of six (6) weeks of once daily application of Furosemide Topical Gel 0.125% (CLS006) compared to vehicle in subjects ≥ 2 years of age with nongenital cutaneous common warts (verruca vulgaris).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have 1 to 6 clearly identifiable common warts located on hands, feet, limbs, and/or trunk

  * Each wart must measure 3 to 10 mm in their longest dimension (diameter) on the epidermal plane of the skin at the baseline visit,
  * Each wart must be present for at least 4 weeks at the baseline visit,
  * Plantar, facial, subungual, and other warts (e.g., flat, genital) are excluded from treatment (i.e., these wart types are excluded from treatment, however the subject is not excluded).
* Male or female subjects 2 years of age or older
* Females of childbearing potential who are using a highly effective form of birth control or females of non-childbearing potential
* Negative in-office urine pregnancy test at Screening and Baseline
* Subjects free of any clinically significant dermatologic disorder in the treatment area
* Subjects free of any clinically significant systemic condition which will interfere with the study assessments or increase the risk of AEs
* Subjects willing to refrain from using other topical products in the treatment area, or prohibited medications for the duration of the study

Exclusion Criteria:

* Subjects who have used any wart treatments/therapies, prescription or over-the-counter, as follows:

  * Salicylic acid, cantharidin, sinecatechins (VeregenTM), simple occlusion (e.g., duct tape), and/or any other over-the-counter wart-removing products in the treatment area within 4 weeks of the Baseline Visit.
  * Cryotherapy (e.g., treatment with liquid nitrogen), carbon dioxide, electrodessication, laser, surgery, or other forms of mechanical destruction (e.g., emery boards, clippers, debriders, etc.) in the treatment area within 8 weeks of the Baseline Visit.
  * Treatment with immunotherapy (DPCP, DNCB or other), imiquimod, 5-fluorouracil, bleomycin, podophyllin or any other wart immunotherapy or treatment (e.g., Candida antigen) designed to stimulate immune response within 12 weeks of the Baseline Visit.
* Female subjects who are pregnant, nursing/breastfeeding, or plan to become pregnant within the study period including the follow-up period.
* Subjects who are immunocompromised.
* Subjects who have taken, within 30 days prior to the Baseline visit, or require treatment with systemic immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) during the course of the study.
* Subjects who require ongoing treatment with oral or injectable furosemide.
* Subjects who have used an investigational drug/device within 30 days of the Baseline visit
* Subjects with known sensitivities to any of the investigational product ingredients including furosemide (or other sulfonamides).
* Subjects with clinically relevant/significant abnormal laboratory results, vital signs, ECG, and/or physical findings at Screening and/or Baseline
* Subjects with a chronic medical condition or clinically significant abnormal physical or laboratory finding(s) that may require the use of a prohibited medication/treatment.
* Subjects who currently abuse alcohol or drugs or who have a history of chronic alcohol or drug abuse within the past year.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Dermatology Specialists, Inc., Oceanside, California
  - West Dermatology Research Center, San Diego, California
  - TCR Medical Corporation, San Diego, California
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - Skin Care Research, Inc., Boca Raton, Florida
  - Dermatology Associates & Research, Coral Gables, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - International Clinical Research - US, LLC, Sanford, Florida
  - Marietta Dermatology Clinical Research, Inc., Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DS Research, New Albany, Indiana
  - Center for Pharmaceutical Research, LLC, Kansas City, Missouri
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - The Dermatology Group, P.C., Verona, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Skin Specialty Dermatology, New York, New York
  - Darst Dermatology, Charlotte, North Carolina
  - Dermatology Specialists of Charlotte, Charlotte, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Oregon Dermatology And Research Center, Portland, Oregon
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - PEAK Research, LLC, Upper Saint Clair, Pennsylvania
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Palmetto Clinical Trial Services, LLC, Fountain Inn, South Carolina
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Arlington Research Center, Inc., Arlington, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Austin Institute for Clinical Research, Inc, Pflugerville, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects must have 1 to 6 clearly identifiable common warts located on hands, feet, limbs, and/or trunk
Groups:
- CLS006: Furosemide Topical Gel applied once daily Furosemide Topical Gel, 0.125%
- CLS006 Vehicle: Vehicle Topical Gel applied once daily Vehicle Topical Gel
Period: Overall Study
Arm/Group | CLS006 | CLS006 Vehicle
Started | 245 | 246
Subjects Who Had 1 Wart | 112 | 118
Subjects Who Had 2 Warts | 48 | 40
Subjects Who Had 3 Warts | 25 | 31
Subjects Who Had 4 Warts | 13 | 18
Subjects Who Had 5 Warts | 20 | 20
Subjects Who Had 6 Warts | 27 | 19
Completed | 226 | 217
Not Completed | 19 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLS006 | CLS006 Vehicle | Total
Number analyzed (Participants) | 245 | 246 | 491
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (18.80) | 30.2 (17.26) | 31.1 (18.05)
Age, Customized [Count of Participants; unit: Participants]
  >=2 to <12 | 39 | 41 | 80
  >=12 to <18 | 40 | 40 | 80
  >=18 to <65 | 150 | 157 | 307
  >=65 | 16 | 8 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 129 | 267
  Male | 107 | 117 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 69 | 116
  Not Hispanic or Latino | 198 | 177 | 375
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 8 | 9 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 5 | 11 | 16
  White | 219 | 211 | 430
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Difference in the Proportion of Subjects With Complete Clearance of All Treated Warts Between the Active and Vehicle at Week 18/End of Post-treatment Efficacy Evaluation
Time Frame: Week 18
Measure: Count of Participants; unit: Participants
Arm/Group | CLS006 | CLS006 Vehicle
Number analyzed (Participants) | 226 | 217
Participants
  Achieved complete clearance of all treated warts | 35 | 27
  Not achieved complete clearance of all treated warts | 191 | 190
Statistical Analysis 1: Comparison: CLS006; Test type: Superiority; p = 0.2587, Cochran-Mantel-Haenszel

2. Secondary Outcome: The Ratio of the Number of Cleared Warts Out of the Number of Treated Warts for Each Subject
Time Frame: Week 18
Measure: Mean (Standard Deviation); unit: Ratio of Cleared Warts
Arm/Group | CLS006 | CLS006 Vehicle
Number analyzed (Participants) | 226 | 217
Ratio of Cleared Warts | 0.210 (0.3771) | 0.191 (0.3500)

3. Secondary Outcome: Difference in the Proportion of Subjects With Complete Clearance of All Treated Warts at Week 12
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | CLS006 | CLS006 Vehicle
Number analyzed (Participants) | 226 | 217
Participants
  Complete clearance of all treated warts | 21 | 19
  Not complete clearance of all treated warts | 205 | 198

4. Secondary Outcome: The Ratio of the Number of Cleared Warts Out of the Number of Treated Warts for Each Subject at Week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: ratio of cleared warts
Arm/Group | CLS006 | CLS006 Vehicle
Number analyzed (Participants) | 226 | 217
ratio of cleared warts | 0.135 (0.3112) | 0.127 (0.3020)

5. Secondary Outcome: Change From Baseline in Wart Size for Each Subject
Time Frame: Week 18
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CLS006 | CLS006 Vehicle
Number analyzed (Participants) | 226 | 217
mm | -3.5 (7.10) | -3.1 (6.84)

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | CLS006 | CLS006 Vehicle
All-Cause Mortality (participants affected / at risk) | 1/245 | 1/246
Serious Adverse Events (participants affected / at risk) | 3/245 | 3/246
Other Adverse Events (participants affected / at risk) | 23/245 | 14/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLS006 (N=245) | CLS006 Vehicle (N=246)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bacterial colitis (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CLS006 (N=245) | CLS006 Vehicle (N=246)
Nausea (Gastrointestinal disorders) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 4
Nasopharyngitis (Infections and infestations) | 4 | 3
Influenza (Infections and infestations) | 3 | 2
Pharyngitis streptococcal (Infections and infestations) | 3 | 2
Sinusitis (Infections and infestations) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT03259620/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT03259620/SAP_001.pdf